CLINICAL TRIAL: NCT02198677
Title: Randomized Trial of Cardiovascular Response to Two Manual Techniques Non-thrust Joint Manipulation of the Cervical Spine in Patients With Non-traumatic Mechanical Neck Pain.
Brief Title: Cardiovascular Response to Two Manual Techniques for Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azusa Pacific University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP vs LAT
Record Dates: First submitted 2014-07-15; First posted 2014-07-24 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AP (Experimental): Anterior to posterior pressures 5x10 seconds per set with 10 seconds rest between each set
  Interventions: Procedure: Anterior to posterior pressures
- Lateral glides (Experimental): Lateral glides 5x10 seconds per set with 10 seconds rest between each set
  Interventions: Procedure: Lateral glide

INTERVENTIONS:
Procedure: Anterior to posterior pressures — Anterior to posterior pressures
  Arms: AP
Procedure: Lateral glide — Lateral glide
  Arms: Lateral glides

SUMMARY:
The aim of the investigators study is to investigate whether posteriorly directed (AP) pressures and laterally directed (LAT) glides, cause blood pressure and heart rate elevation or lowering in patients with neck pain. The answer will advance the investigators understanding of why manual therapy works.

DETAILED DESCRIPTION:
To be included in the study, these subjects with unilateral non-traumatic, non-chronic neck pain (operationally defined as neck pain with mobility deficits lasting less than 3 months) shall have numeric pain rating scale (NPRS) of between 0 and 5 out of 10 as the most painful neck movement even with passive scapular elevation, neck disability index (NDI) of between 16 and 50 out of 100%, resting systolic and diastolic blood pressure between 90/60 and 138/88, and resting heart rate between 60 and 90. Subjects are excluded if they are current smoker, over 50 years of age, has a history of fainting spells or loss of consciousness, is on blood thinners, is taking medications for or have a history of diabetes mellitus, neurologic or cardiovascular disease, has a history of spinal surgeries, and has neck pain classified or associated with headache, radiating pain, and movement coordination impairments. A convenience sample of subjects will be randomly allocated to 1 of 2 groups. Both Group 1: AP and Group 2: LAT will receive posterior pressures and lateral glides respectively to one hypomobile segment. Baseline NPRS, and NDI will be collected at the initial visit. Systolic blood pressure (SBP) and heart rate (HR) will be measured with a OMRON automatic monitor recording time points: (1) 5 minutes, and (2) 7 minutes after lying supine; (3) during the 1st set, (4) 5th set of one of the glides, (5) 2 minutes after time point #4, and (6) 4 minutes after time point #4. After time point #6, a global rating of change (GROC) will immediately be collected based on the most painful neck movement. A finger pulse oximeter will be placed on the subjects' index finger to constantly monitor their pulse rate for slowing heart rate or asystole. The primary author will perform one of the techniques on all subjects. After one visit, a follow-up NPRS, and NDI will be collected again.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral, non-traumatic, non-chronic mechanical neck pain
* Numeric pain rating scale between 0-5/10 as the most painful neck movement (with passive scapular elevation)
* Neck Disability Index between 16-50/100 percent
* Resting blood pressure between 90/60 and 138/88 mmHg
* Resting heart rate between 60 and 90 beats per minute

Exclusion Criteria:

* Current smoker
* Under 18 years and over 50 years of age
* History of fainting spells or loss of consciousness
* Currently on blood thinners
* Taking medications for or have a history of diabetes mellitus, neurologic or cardiovascular disease
* History of spinal surgery
* Has neck pain classified or associated headache, arm pain, trauma/whiplash

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate | 7 minutes before, 5 minutes before, During first set, During fifth set, 2 minutes after time point 4, 4 minutes after time point 4

SECONDARY OUTCOMES:
Change in blood pressure | 7 minutes before, 5 minutes before, During first set, During fifth set, 2 minutes after time point 4, 4 minutes after time point 4
Change in Numeric Pain Rating Scale | Baseline and within 7 days after the intervention
Change in Neck Disability Index | Baseline and 7 days after the intervention
Global rating of change | Immediately after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wong, DPT, Principal Investigator — Azusa Pacific University; Emmanuel Yung, DPT, Principal Investigator — Sacred Heart University
Locations (1):
- Physical Therapy Department, Azusa, California, United States

REFERENCES:
- [Background] Childs JD, Cleland JA, Elliott JM, Teyhen DS, Wainner RS, Whitman JM, Sopky BJ, Godges JJ, Flynn TW; American Physical Therapy Association. Neck pain: Clinical practice guidelines linked to the International Classification of Functioning, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2008 Sep;38(9):A1-A34. doi: 10.2519/jospt.2008.0303. Epub 2008 Sep 1. PMID 18758050
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Result] Bruehl S, Dengler-Crish CM, Smith CA, Walker LS. Hypoalgesia related to elevated resting blood pressure is absent in adolescents and young adults with a history of functional abdominal pain. Pain. 2010 Apr;149(1):57-63. doi: 10.1016/j.pain.2010.01.009. Epub 2010 Feb 1. PMID 20122805
- [Result] Hurwitz EL, Morgenstern H, Vassilaki M, Chiang LM. Frequency and clinical predictors of adverse reactions to chiropractic care in the UCLA neck pain study. Spine (Phila Pa 1976). 2005 Jul 1;30(13):1477-84. doi: 10.1097/01.brs.0000167821.39373.c1. PMID 15990659
- [Result] Knutson GA. Significant changes in systolic blood pressure post vectored upper cervical adjustment vs resting control groups: a possible effect of the cervicosympathetic and/or pressor reflex. J Manipulative Physiol Ther. 2001 Feb;24(2):101-9. doi: 10.1067/mmt.2001.112564. PMID 11208222
- [Result] Krediet CT, Jardine DL, Wieling W. Dissection of carotid sinus hypersensitivity: the timing of vagal and vasodepressor effects and the effect of body position. Clin Sci (Lond). 2011 Nov;121(9):389-96. doi: 10.1042/CS20100607. PMID 21595633
- [Result] Lidegaard O, Lokkegaard E, Jensen A, Skovlund CW, Keiding N. Thrombotic stroke and myocardial infarction with hormonal contraception. N Engl J Med. 2012 Jun 14;366(24):2257-66. doi: 10.1056/NEJMoa1111840. PMID 22693997
- [Result] Lidegaard O, Nielsen LH, Skovlund CW, Skjeldestad FE, Lokkegaard E. Risk of venous thromboembolism from use of oral contraceptives containing different progestogens and oestrogen doses: Danish cohort study, 2001-9. BMJ. 2011 Oct 25;343:d6423. doi: 10.1136/bmj.d6423. PMID 22027398
- [Result] McGuiness J, Vicenzino B, Wright A. Influence of a cervical mobilization technique on respiratory and cardiovascular function. Man Ther. 1997 Nov;2(4):216-220. doi: 10.1054/math.1997.0302. PMID 11440535
- [Result] Puentedura EJ, Cleland JA, Landers MR, Mintken PE, Louw A, Fernandez-de-Las-Penas C. Development of a clinical prediction rule to identify patients with neck pain likely to benefit from thrust joint manipulation to the cervical spine. J Orthop Sports Phys Ther. 2012 Jul;42(7):577-92. doi: 10.2519/jospt.2012.4243. Epub 2012 May 14. PMID 22585595
- [Result] Van Dillen LR, McDonnell MK, Susco TM, Sahrmann SA. The immediate effect of passive scapular elevation on symptoms with active neck rotation in patients with neck pain. Clin J Pain. 2007 Oct;23(8):641-7. doi: 10.1097/AJP.0b013e318125c5b6. PMID 17885341
- [Result] Egwu MO. Relative therapeutic efficacy of some vertebral mobilization techniques in the management of unilateral cervical spondylosis: a comparative study. Journal of Physical Therapy and Science. 2008;20:103-8.